CLINICAL TRIAL: NCT04110951
Title: The Effect of Pranayama Breathing Technique on Asthma Control, Pulmonary Function and Quality of Life: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Pranayama Breathing Technique on Asthma Control, Pulmonary Function and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gülyeter Erdoğan Yüce, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2017-7652
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: Asthma; Yoga; Breathing exercises; Quality of life; Nursing
MeSH Terms: conditions — Asthma | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama group (Experimental): Kapalbhati, Ujjayi and Anuloma-Viloma pranayama techniques were applied to the experimental group. Within this scope, a three days of applied training program was prepared and a guide involving the steps of Pranayama breathing technique was formed. The patients in of pranayama group were trained by the researcher who had yoga trainer certificate. After completing three days of training and observations regarding their accomplishment of applications properly, a pranayama breathing technique video showing how the pranayama breathing technique is done with its details was downloaded to their smartphones and a guide including the application steps was distributed to the patients. The patients were required to apply pranayama technique, in company with the video, 20 min every day and a month in total.
  Interventions: Behavioral: Pranayama Breathing Technique
- Relaxation group (Active Comparator): As there was not placebo breathing control treatment appropriate to yoga breathing technique, relaxation technique was decided to apply in the second group to equalize psychological effects of the treatment. Progressive relaxation technique was taught to the relaxation group during the same training span.A three days of applied training program and Relaxation Technique Application Guide, including steps of progressive relaxation technique, were prepared within this scope. After completing three days of training and observations regarding their accomplishment of applications properly, a relaxing music to listen during applications and a training video involving progressive relaxation directives were downloaded to smartphones of the patients. Also, Relaxation Technique Application Guide involving application steps were distributed to the patients. The patients were required to apply relaxation technique, in company with the video, 20 min every day and a month in total.
  Interventions: Behavioral: Relaxation technique

INTERVENTIONS:
Behavioral: Pranayama Breathing Technique — Yogic Breathing Technique
  Arms: Pranayama group
Behavioral: Relaxation technique — Progressive relaxation technique
  Arms: Relaxation group

SUMMARY:
Most of the asthma patients prefer complementary and integrative applications as they continue to experience asthma symptoms despite pharmacological treatment. Pranayama, one of these treatments, is a breathing-based technique and is a part of yoga, an ancient Indian science. This study was carried out as randomized controlled single blind study in order to analyze the effect of pranayama breathing technique applied to individuals suffering from asthma on asthma control, pulmonary functions and quality of life. The study comprised 50 patients in total, as 25 patients in pranayama group and 25 patients in control group. The approval of ethics committee, permissions from the institutions, and informed voluntary approval of the individuals were obtained to conduct the research. The data of the research were collected through the application of Asthma Control Test (ACT), Asthma Quality of Life Questionnaire (AQLQ), pulmonary function test (PFT), and patient observation chart. Pranayama breathing technique was applied to pranayama group 20 minutes once a day for four weeks, and relaxation technique was applied to relaxation group similarly in addition to standard treatment. ACT, AQLQ, and PFT were evaluated twice as before and after the one month of application process. Meanwhile, the patients' PEF measurements were followed with individual PEF meter on daily basis. The value of p<0.05 was accepted statistically significant in the data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Can communicate,
* To have an increase of %12 or 200 ml in FEV1 value after inhaler bronchodilator at breathing function test,
* To have chronic asthma diagnose with 6 months approved by doctors and receiving treatment,
* Asthma controls are not under control or partly under control in relation to GINA (Global Initiative for Asthma) values,
* Taking beta2-agonist and/or ICS twice a week or more to control asthma symptoms,
* There is not any chance in inhaler bronchodilator drug potions during the last four weeks,
* Can use a smart phone.

Exclusion Criteria:

* To have lung diseases such as COPD,
* To have tuberculosis and respiratory infection,
* To have diabetes and coronary artery disease,
* Smokers
* Pregnant or nursing mother,
* Doing regular exercise,
* Benefitng from other complementary and integrative health applications during treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test | change from baseline score at the end of one month
  Asthma Control Test (ACT) is composed of 5 main sections involving asthma influence level of patients due to daily actions of patients, frequency of asthma symptoms at daytimes and nights, need of urgent relaxing drug, and evaluation of disease by patients. Patients are required to respond each question with values between 1 and 5. Total score of these 5 questions ranges between 5 and 25
Asthma Quality of Life Questionnaire | change from baseline score at the end of one month
  Standard Asthma Quality of Life Questionnaire (AQLQ) is a quality of life questionnaire specific to asthma comprising 32 questions. AQLQ was developed by Juniper et al. (1993) to use in clinical studies. The questionnaire evaluates responses through a 7 scores scale (1: severely impaired; 7: not impaired at all) based on changes in last two weeks regarding asthma. Standard AQLQ involves 12 questions about symptoms, 11 questions about activity limitation, 5 questions about emotional functions, and 4 questions about environment stimuli. Mean scores are calculated for subcategories and overall scores. The mean of obtained scores are evaluated between 1 and 7. The minimum score change clinically accepted important in the questionnaire is 0.50 and this situation is called "minimal significant difference" .
Peak Ekspiratuar Flow | change from baseline score at the end of one month
  Peak Ekspiratuar Flow (PEF) measurement kind of test which can be accomplished through mobile hand-held tools that enable patients to follow their situations even at their own homes in asthma diagnose and treatment. Repeatability of the test is very high though its application is connected with effort. As PEF measurement gives information about big airways, lower values are obtained in comparison to FEV1 value at 30-50% of the patients. In PEF follow-up, the best PEF value of patient value is primarily defined. Because, the follow-up of patient is conducted in terms of his/her best value not in terms of prediction value indifferent to spirometer in PEF follow-up.
Forced Expiratory Volume First Second | change from baseline score at the end of one month
  Forced expiratory volume in first second (FEV1), measured during breathing function test and a flow velocity, is the best indicator of obstruction in asthma. However, FEV1 reflects real obstruction only with powerful and maximum effort as it mostly related with effort.
Forced Vital Capacity | change from baseline score at the end of one month
  Effort related part of forced vital capacity (FVC) reflects airways, pulmonary expriratory muscles and the situation of lung elastic recession power.
FEV1/FVC | change from baseline score at the end of one month
  FEV1/FVC rate is an important final parameter in defining obstruction as there is not a great change observed in FVC values at early stages of the disease in most of the asthma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevşehir Haci Bektaş Veli Üniversitesi, Nevşehir, Nerkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans.

REFERENCES:
- [Background] Agarwal D, Gupta PP, Sood S. Assessment for Efficacy of Additional Breathing Exercises Over Improvement in Health Impairment Due to Asthma Assessed using St. George's Respiratory Questionnaire. Int J Yoga. 2017 Sep-Dec;10(3):145-151. doi: 10.4103/0973-6131.213472. PMID 29422745
- [Background] Aggarwal T, Khatri A, Siddiqui SS, Hasan SN, Singh D, Kulshreshtha M, Agarwal S. Pranayama has additive beneficial effects along with medication in bronchial asthma patients. Journal of Physiology and Pharmacology Advances, 2013; 3(12): 292-297.
- [Background] Agnihotri S, Kant S, Mishra SK, Verma A. Assessment of significance of Yoga on quality of life in asthma patients: A randomized controlled study. Ayu. 2017 Jan-Jun;38(1-2):28-32. doi: 10.4103/ayu.AYU_3_16. PMID 29861589
- [Background] Arulmozhi S, Joice SP, Maruthy KN. Effect of pranayama on respiratory muscle strength in chronic asthmatics. National Journal of Physiology, Pharmacy and Pharmacology, 2018; 8(12): 1700-1703.
- [Background] Bhatt A, Rampallivar S. Effect of pranayam on ventilatory functions in patients of bronchial asthma. Journal of evolution of medical and dental sciences-jemds, 2016; 5(28): 1453-1455.
- [Background] Cooper S, Oborne J, Newton S, Harrison V, Thompson Coon J, Lewis S, Tattersfield A. Effect of two breathing exercises (Buteyko and pranayama) in asthma: a randomised controlled trial. Thorax. 2003 Aug;58(8):674-9. doi: 10.1136/thorax.58.8.674. PMID 12885982
- [Background] Cowie RL, Conley DP, Underwood MF, Reader PG. A randomised controlled trial of the Buteyko technique as an adjunct to conventional management of asthma. Respir Med. 2008 May;102(5):726-32. doi: 10.1016/j.rmed.2007.12.012. Epub 2008 Jan 31. PMID 18249107
- [Background] Fluge T, Richter J, Fabel H, Zysno E, Weller E, Wagner TO. [Long-term effects of breathing exercises and yoga in patients with bronchial asthma]. Pneumologie. 1994 Jul;48(7):484-90. German. PMID 7937658
- [Background] George M, Topaz M. A systematic review of complementary and alternative medicine for asthma self-management. Nurs Clin North Am. 2013 Mar;48(1):53-149. doi: 10.1016/j.cnur.2012.11.002. Epub 2013 Jan 10. PMID 23465447
- [Background] Gulati K, Babita R. A clinical study to evaluate the effects of yogic intervention on pulmonary functions, inflammatory markers and quality of life in patients of bronchial asthma. EC Pharmacology and Toxicology, 2017; 3: 174-181.
- [Background] Hoang KAT, Nguyen HM. The effectiveness of practicing pranayama yoga on some respiratory indicators in patients suffering from bronchial disease. International Journal of Science Culture and Sport (IntJSCS), 2015; 3(2): 6-12.
- [Background] Holloway EA, West RJ. Integrated breathing and relaxation training (the Papworth method) for adults with asthma in primary care: a randomised controlled trial. Thorax. 2007 Dec;62(12):1039-42. doi: 10.1136/thx.2006.076430. Epub 2007 Jun 15. PMID 17573445
- [Background] Husseın NA, Afıfy AM, Obaya HE, Rafea AS. Effects of Ujjayi Pranayama Trainning on Selected Ventilatory Function Test in Patients with Mild Bronchial Asthma. Med. J. Cairo Univ., 2016; 84(2): 445-452.
- [Background] Jerath R, Edry JW, Barnes VA, Jerath V. Physiology of long pranayamic breathing: neural respiratory elements may provide a mechanism that explains how slow deep breathing shifts the autonomic nervous system. Med Hypotheses. 2006;67(3):566-71. doi: 10.1016/j.mehy.2006.02.042. Epub 2006 Apr 18. PMID 16624497
- [Background] Kant S, Agnihotri S. Asthma diagnosis and treatment-1029. Yoga as an adjuvant therapy in asthma management. In World Allergy Organization Journal, 2013; 6(1): 28.
- [Background] Karam M, Kaur BP, Baptist AP. A modified breathing exercise program for asthma is easy to perform and effective. J Asthma. 2017 Mar;54(2):217-222. doi: 10.1080/02770903.2016.1196368. Epub 2016 Jun 10. PMID 27285510
- [Background] Karmakar S, Karmakar S. The Role of Yoga in Bronchial Asthma. J Complement Med Alt Healthc. J, 2018; 7(2): 1-4.
- [Background] Malarvizhi M, Maheshkumar K. Effect of 6 months of yoga practice on quality of life among patient with asthma: a randomized control trial. Advances in Integrative Medicine, 2018, 1-8.
- [Background] Manivannan D. Effect of Yoga Therapy on Clinical Profile and PEFR among Women with Bronchial Asthma. Indian Journal of Ancient Medicine and Yoga, 2017; 10(4): 125-130.
- [Background] Manocha R, Marks GB, Kenchington P, Peters D, Salome CM. Sahaja yoga in the management of moderate to severe asthma: a randomised controlled trial. Thorax. 2002 Feb;57(2):110-5. doi: 10.1136/thorax.57.2.110. PMID 11828038
- [Background] Morse D. Yoga for asthma. International Journal of Yoga Therapy, 2007; 17(1): 81-88. Morse, 2007
- [Background] Murthy KJ, Sahay BK, Sitaramaraju P, Sunita M, Yogi R, Annapurna N, Ramesh M, Prasad V, Reddy E. Effect of pranayama (rechaka, puraka and kumbaka) on bronchial asthma-an open study. Lung India, 1984; 2(2): 187-191.
- [Background] Nagarathna R, Nagendra HR. Yoga for bronchial asthma: a controlled study. Br Med J (Clin Res Ed). 1985 Oct 19;291(6502):1077-9. doi: 10.1136/bmj.291.6502.1077. PMID 3931802
- [Background] Prem V, Sahoo RC, Adhikari P. Comparison of the effects of Buteyko and pranayama breathing techniques on quality of life in patients with asthma - a randomized controlled trial. Clin Rehabil. 2013 Feb;27(2):133-41. doi: 10.1177/0269215512450521. Epub 2012 Jul 26. PMID 22837543
- [Background] Pandit DP, Vaidya SM. Effect of yoga on pulmonary function tests in patients of bronchial asthma. International Journal 2013; 2(3): 58-63.